CLINICAL TRIAL: NCT05261334
Title: Socket Shielding in Immediate Versus Early Implant Placement With Contour Augmentation of Fresh Extraction Sockets in the Esthetic Zone. A Randomized Pilot Clinical Study.
Brief Title: Socket Shield Technique Versus Early Implant Placement With Contour Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Iman Abd-ElWahab Radi, PhD (Other)
Responsible Party: Sponsor-Investigator, Iman Abd-ElWahab Radi, PhD, Professor of Prosthodontics, Faculty of Dentistry, Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sst versus contour aug
Record Dates: First submitted 2022-01-28; First posted 2022-03-02 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Bone Loss; Bone Resorption
MeSH Terms: conditions — Bone Diseases, Metabolic; Bone Resorption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- socket shield technique (Active Comparator): immediate implant placement with socket shield technique
  Interventions: Procedure: contour augmentation
- contour augmentation (Active Comparator): early implant placement with contour bone augmentation
  Interventions: Procedure: contour augmentation

INTERVENTIONS:
Procedure: contour augmentation — early implant placement with contour bone augmentation

SUMMARY:
comparing socket shield technique with early implant placement with contour augmentation in preserving the bone contour

DETAILED DESCRIPTION:
comparing immediate implant placement with socket shield technique and final crown after 3 months with extraction and after 4 to 8 weeks implant placement with contour bone augmentation then after 3 to 4 months final crown delivery

ELIGIBILITY:
Inclusion Criteria:

1. Non-restorable maxillary teeth in the esthetic zone
2. Intact adjacent teeth
3. Adequate palatal and apical bone that allows achieving implant primary stability.
4. Type I socket
5. ≥18 years
6. ≤ 60 years
7. Systemically healthy patients

Exclusion Criteria:

1. Extraction sockets with acute or chronic infection or with adjacent infected teeth
2. Heavy Smokers > than 10 cigarettes daily
3. Cancer patients undergoing radiotherapy or chemotherapy during or within the last 6 months.
4. Unmotivated patients to maintain adequate oral hygiene to follow up.
5. Patients with physical disabilities that could affect follow up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-31 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
facial bone thickness | 12 months
  using superimposed CBCT images

SECONDARY OUTCOMES:
facial bone height changes | 12 months
  using superimposed CBCT images
Soft tissue height changes | 12 months
  using superimposed intraoral scans

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided